CLINICAL TRIAL: NCT00055419
Title: A Phase II Study of Cetuximab in Patients Who Have Stage IV Colorectal Cancer
Brief Title: A Study of Cetuximab in Patients Who Have Stage IV Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-041
Record Dates: First submitted 2003-02-28; First posted 2003-03-04 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Colorectal Neoplasms
Keywords: Stage IV colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 400 mg/m2 (Experimental)
  Interventions: Biological: Cetuximab

INTERVENTIONS:
Biological: Cetuximab — 400 mg/m2 loading dose Week 1, followed by 250 mg/m2 weekly until disease progression
  Other Names: Erbitux

SUMMARY:
The purpose of this clinical research study is to learn about the safety of cetuximab in patients with stage IV colorectal cancer, and who may benefit from cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed an approved informed consent prior to any study procedures.
* Subjects with histologically or pathologically confirmed metastatic colorectal cancer, which is EGFR-positive by IHC (may be based on archival samples)
* Subjects with ECOG performance status 0, 1 or 2.
* Subjects who have failed, either due to lack of efficacy or due to intolerance, all available chemotherapy for the treatment of metastatic colorectal cancer.
* Subjects who have failed to meet eligibility criteria for any other existing cetuximab trial.
* Subjects must have received at least two chemotherapy regimens for metastatic disease OR adjuvant therapy plus one chemotherapy regimen for metastatic disease, provided the subject progressed within 6 months of completing their adjuvant therapy.
* Prior chemotherapy must have included all of the follow drugs: irinotecan, oxaliplatin, and a fluoropyrimidine.
* Subjects adequately recovered from any recent surgery, radiation therapy or chemotherapy.
* Subjects accessible for treatment and follow-up. Subjects enrolled in this trial must be treated at the participating center.
* Subjects greater or equal to 18 years of age.
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks afterwards.

Exclusion Criteria:

* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Sexually active, fertile men not using adequate birth control.
* Subjects with dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Subjects with a serious uncontrolled medical disorder that would impair the ability of the patient to receive protocol therapy.
* Subjects with a history of uncontrolled angina, arrhythmias, congestive heart failure, or myocardial infarction within the previous 6 months.
* Subjects with any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. Subjects with a previous malignancy but without evidence of disease for > 5 years will be allowed to enter the trial.
* Subjects with any history of severe hypersensitivity reactions and/or anaphylaxis resulting from the administration of protein based therapeutic agents.
* Subjects with inadequate hematologic function defined by an absolute neutrophil count (ANC) <1,250/mm3, a platelet count <75,000/mm3, and a hemoglobin level <8 g/dL.
* Subjects with inadequate hepatic function, defined by a total bilirubin level ³3 times the upper limit of normal (ULN) and an aspartate transaminase (AST) and alanine transaminase (ALT) levels >5 x ULN.
* Subjects with inadequate renal function defined by a serum creatinine level >2.5 x ULN.
* Prior cetuximab therapy, prior randomization on a study which includes cetuximab therapy in a treatment arm, or any other prior therapy that targets the EGFR pathway.
* A history of prior therapy with a chimerized or murine monoclonal antibody.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.
* A history of cetuximab or therapy that targeted the EGFR receptor.
* A history of prior anti-cancer murine monoclonal antibody therapy.
* Additional concurrent chemotherapy or other investigational anticancer agents may not be administered to subjects on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2003-02; Primary Completion 2004-07 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
The objective of this study will be to monitor the safety of administering cetuximab,via an access program, to subjects with metastatic colorectal carcinoma who have exhausted all standard therapies or treatment options. | Every 4 weeks untill disease progression

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (29):
- United States (29):
  - ImClone Investigational Site, Bakersfield, California
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Denver, Colorado
  - ImClone Investigational Site, Torrington, Connecticut
  - ImClone Investigational Site, Washington D.C., District of Columbia
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, Miami, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Decatur, Illinois
  - ImClone Investigational Site, Louisville, Kentucky
  - ImClone Investigational Site, New Orleans, Louisiana
  - ImClone Investigational Site, Baltimore, Maryland
  - ImClone Investigational Site, Ypsilanti, Michigan
  - ImClone Investigational Site, Minneapolis, Minnesota
  - ImClone Investigational Site, Saint Charles, Missouri
  - ImClone Investigational Site, Great Falls, Montana
  - ImClone Investigational Site, Las Vegas, Nevada
  - ImClone Investigational Site, Voorhees Township, New Jersey
  - ImClone Investigational Site, East Setauket, New York
  - ImClone Investigational Site, Latham, New York
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Cleveland, Ohio
  - ImClone Investigational Site, Portland, Oregon
  - ImClone Investigational Site, Greenville, South Carolina
  - ImClone Investigational Site, Memphis, Tennessee
  - ImClone Investigational Site, Dallas, Texas
  - ImClone Investigational Site, Norfolk, Virginia
  - ImClone Investigational Site, Green Bay, Wisconsin